CLINICAL TRIAL: NCT01208168
Title: A Randomized, Double-Blind, Vehicle-Controlled, Multicenter, Parallel Group Study of the Safety and Efficacy of NAB001 in the Treatment of Mild to Moderate Distal Subungual Onychomycosis of the Toenails for 52 Wks
Brief Title: Safety & Efficacy of NAB001 in the Treatment of Mild to Moderate Onychomycosis of the Toenails
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Promius Pharma, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0904
Record Dates: First submitted 2010-09-20; First posted 2010-09-23 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Onychomycosis
Keywords: toenail fungus; onychomycosis; nail infection
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active drug (Experimental)
  Interventions: Drug: NAB001
- Vehicle alone (Placebo Comparator)
  Interventions: Drug: Vehicle alone

INTERVENTIONS:
Drug: NAB001 — nail lacquer, once daily, 52 weeks
  Arms: Active drug
Drug: Vehicle alone — nail lacquer, once daily, 52 weeks
  Arms: Vehicle alone

SUMMARY:
The objectives of this study are to assess the safety of NAB001 for topical treatment of mild to moderate distal onychomycosis of the toenails over 52 weeks and to compare the efficacy of NAB001 to vehicle alone at the end of the study (Week 56) after treating for 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* mild to moderate fungal infection of the toenail as assessed by study doctor
* koh positive & dermatophyte culture positive at Visit 1
* good general health as assessed by the study doctor

Exclusion Criteria:

* severe fungal toenail infection
* prior use of antifungal drugs (wash-out allowed, duration varies on class)
* significant confounding conditions as assessed by study doctor
* pregnancy/lactation
* must forego nail salon procedures during study for at least ~60 weeks

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Actual)
Dates: Start 2010-09; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Complete cure rate at Week 56. Complete cure defined as clinically clear nail and mycological cure. | Week 56 after 52 weeks of treatment

SECONDARY OUTCOMES:
Proportion of subjects with effective treatment at week 56. Effective treatment defined as mycological cure and an IGA of 0 or 1 (Clear or almost clear). | Week 56

CONTACTS AND LOCATIONS:
Overall Officials: Kent Allenby, MD, Study Director — Promius Pharma; Joanne Fraser, PhD, Study Director — Promius Pharma
Locations (24):
- United States (22):
  - Phoenix, Arkansas
  - T. Joseph Raoof, MD, Inc., Encino, California
  - Skin Surgery Medical Group, Inc., San Diego, California
  - Longmont Medical Research Network, Longmont, Colorado
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Internaional Dermatology Research, Inc., Miami, Florida
  - MedaPhase, Inc., Newnan, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Northwest Clinical Trials, Boise, Idaho
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Gerard Furst, DPM, PLLC, East Setauket, New York
  - Dermatology Consulting Services, High Point, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Mazur Foot and Ankle, Salisbury, North Carolina
  - Radiant Research, Cincinnati, Ohio
  - Oregon Dermatology & Research Network, Portland, Oregon
  - Temple University - School of Podiatric Medicine, Philadelphia, Pennsylvania
  - Carolina Dermatology of Greenville, PA, Greenville, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - Ashton Podiatry Associates, PA, Dallas, Texas
  - Progressive Clinical Research, San Antonio, Texas
- Dominican Republic (2):
  - Instituto Dermatologica, Santo Domingo
  - Instituto Dermatologico, Santo Domingo